CLINICAL TRIAL: NCT07300904
Title: A Randomized, Controlled, Blinded, Prospective, Multi-center Study Evaluating Tensi+ With Transcutaneous Tibial Nerve Stimulation for the Treatment of Overactive Bladder Syndrome
Brief Title: Tensi+ for Treating Overactive Bladder: A Randomized Controlled Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stimuli Technology (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CIP-PF0001-02
Record Dates: First submitted 2025-12-21; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Overactive Bladder (OAB)
Keywords: Overactive Bladder; Transcutaneous Tibial Nerve Stimulation; Urology
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Tensi+ device to be delivered for use by patient (Active Comparator)
  Interventions: Device: Tensi+
- Identical Tensi+ Sham device to be delivered for use by patient (Sham Comparator)
  Interventions: Device: Tensi+

INTERVENTIONS:
Device: Tensi+ — Transcutaneous Tibial Nerve Stimulation

SUMMARY:
The purpose of the study is to evaluate the safety and effectiveness of the Tensi+ device using Transcutaneous Posterior Tibial Nerve Stimulation (TPTNS) for treating patients suffering from OAB symptoms urinary frequency, urgency, with or without urge urinary incontinence.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects aged 22 years or older and,
* Diagnosed with OAB symptoms (characterized by urinary urgency, with or without UUI),
* Symptoms persisting for at least 3 months, and
* Documented with 2 or more urgency episodes per day (with or without incontinence) in two 3-day bladder diaries and,
* With at least 11 or more voids per day (urinary frequency) documented in two 3-day bladder diaries
* Willing and capable of providing informed consent
* Capable of participating in all testing associated with this clinical investigation

Exclusion Criteria:

* Patients with pacemakers or implanted defibrillators or any other implanted electronic device
* Patients prone to excessive bleeding
* Patients with nerve damage that could impact the percutaneous tibial nerve or pelvic floor function
* Patients who are pregnant or planning to become pregnant while using this product
* Patients with ankle joint problems, ankle oedema or dermatological oedema in the area where the electrodes should be placed
* Patients wearing a metal implant near the stimulated area
* Patient with cognitive deficiency
* Administration of intravesical injection of botulinum toxin within 12 months of study enrollment, or treatment within the previous year with other forms neuromodulation for OAB
* Patients treated with medical therapy OAB treatment washout inferior to 30 days
* Patients with diabetic neuropathy
* Patients with uncontrolled diabetes and HbA1c levels above 7%
* Guillain-Barré syndrome
* Chronic inflammatory demyelinating polyneuropathy (CIDP)
* Multiple sclerosis
* A primary diagnosis of stress urinary incontinence (SUI)
* Patients with recurrent rrinary tract infections (UTIs) defined as more than 2 episodes per year, or with any baseline lower urinary tract pathology identified at the time of the 3-day bladder diary assessment.
* Currently participating in another clinical trial

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Treatment success | 12 weeks
  Percentage of responders in urgency events, where a responder is defined as a subject that either achieves a 50% or greater reduction, from baseline to Week 12, in total urgency events per day, or returns to normal (0 events per day) at Week 12. This endpoint will be evaluated through 3-day bladder diaries.

SECONDARY OUTCOMES:
Frequency of urinary voids | 12 weeks
  Percentage of responders in urinary frequency, where a responder is defined as a subject that either achieves a 30% or greater reduction, from baseline to Week 12, in total urinary frequency per day, or returns to normal
Urge urinary incontinence | 12 weeks
  Percentage of responders in urge urinary incontinence, where a responder is defined as a subject that either achieves a 30% or greater reduction, from baseline to Week 12, in total urinary frequency per day, or returns to normal (0 events per day)
Overall Responder Rate Across OAB Symptoms | 12 weeks
  Overall Responder rate defined as the percentage of responders who meet at least the responder criteria in one of the 3 symptoms of OAB, from baseline to Week 12 (urgency, frequency and UUI) from baseline
Quality of life measures | 12 weeks
  Measured using the OAB-q Short Form (SF) questionnaire, which includes 19 questions scored from 1 ("none of the time") to 6 ("all of the time"). The total score ranges from 19 (best QOL) to 114 (worst QOL). A decrease in score from baseline to Week 12 indicates an improvement in quality of life.
Endurance of effect | 24 weeks
  Maintenance of responder status from the primary endpoint (Week 12) through the last follow-up visit without relapse (Week 24), indicating a sustained treatment effect until the end-of-study visit.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (2):
  - Cedars-Sinai, Beverly Hills, California
  - NYU Langone Health, New York, New York
- Toronto Western Hospital, Toronto, Canada

IPD SHARING:
Plan to Share IPD: No